CLINICAL TRIAL: NCT02964962
Title: REPRISE EDGE 29 mm EU Study: REpositionable Percutaneous Replacement of NatIve StEnotic Aortic Valve Through Implantation of LOTUS EDGE 29 mm Valve - Evaluation of Safety and Performance
Brief Title: REPRISE EDGE 29 mm EU Study
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Currently not moving forward with the study
Sponsor: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: S2351
Record Dates: First submitted 2016-11-13; First posted 2016-11-16 (Estimated); Last update posted 2019-07-05 (Actual); Status verified 2019-07

CONDITIONS: Aortic Valve Stenosis
MeSH Terms: conditions — Aortic Valve Stenosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 29 mm LOTUS Edge™ (Experimental)
  Interventions: Device: 29 mm LOTUS Edge™ Valve System

INTERVENTIONS:
Device: 29 mm LOTUS Edge™ Valve System — Transcatheter aortic valve replacement

SUMMARY:
The objective of the REPRISE EDGE 29 mm EU study is to evaluate performance and safety of the 29 mm LOTUS Edge™ Valve System for transcatheter aortic valve replacement (TAVR) in symptomatic subjects with calcific, severe native aortic stenosis who are considered at extreme or high risk for surgical aortic valve replacement (SAVR).

ELIGIBILITY:
Inclusion Criteria:

1. Subject has documented calcific native aortic valve stenosis with an initial aortic valve area (AVA) of ≤1.0 cm2 (or AVA index of ≤0.6 cm2/m2) and either a mean pressure gradient ≥40 mm Hg or a jet velocity ≥4 m/s, as measured by echocardiography and/or invasive hemodynamics.
2. Subject has a documented aortic annulus size of ≥27 mm and ≤29 mm based on the site's assessment of pre-procedure diagnostic imaging (and confirmed by the Case Review Committee [CRC]).
3. Subject has symptomatic aortic valve stenosis with NYHA Functional Class ≥ II.
4. There is agreement by the heart team (which must include a site investigator interventionalist and a site investigator cardiac surgeon) that subject is at high or extreme operative risk for surgical valve replacement (see Note 5 below for definitions of extreme and high risk, the required level of surgical assessment, and CRC confirmation) and that TAVR is appropriate.

   Additionally, subject has at least one of the following:
   * Society of Thoracic Surgeons (STS) score ≥8% -OR-
   * If STS <8, subject has at least one of the following conditions:

     * Hostile chest
     * Porcelain aorta
     * Severe pulmonary hypertension (>60 mmHg)
     * Prior chest radiation therapy
     * Coronary artery bypass graft(s) at risk with re-operation
     * Severe lung disease (need for supplemental oxygen, FEV1 <50% of predicted, DLCO <60%, or other evidence of severe pulmonary dysfunction)
     * Neuromuscular disease that creates risk for mechanical ventilation or rehabilitation after surgical aortic valve replacement
     * Orthopedic disease that creates risk for rehabilitation after surgical aortic valve replacement
     * Childs Class A or B liver disease (subjects with Childs Class C disease are not eligible for inclusion in this trial)
     * Frailty as indicated by at least one of the following: 5-meter walk >6 seconds, Katz ADL score of 3/6 or less, body mass index <21, wheelchair bound, unable to live independently
     * Age ≥90 years
     * Other evidence that subject is at high or extreme risk for surgical valve replacement (CRC must confirm agreement with site heart team that subject meets high or extreme risk definition)

   Note 5: Risk of operative mortality and morbidity must be assessed via an in-person evaluation by a site cardiac surgeon and must be confirmed by the CRC (which must include an experienced cardiac surgeon). Extreme operative risk and high operative risk are defined as follows:

   Extreme Operative Risk: Predicted operative mortality or serious, irreversible morbidity risk ≥50% at 30 days.

   High Operative Risk: Predicted operative mortality or serious, irreversible morbidity risk ≥15% at 30 days.
5. Heart team (which must include a cardiac interventionalist and an experienced cardiac surgeon) agrees that the subject is likely to benefit from valve replacement.
6. Subject (or legal representative) understands the study requirements and the treatment procedures, and provides written informed consent.
7. Subject, family member and/or legal representative agree(s) and subject is capable of returning to the study hospital for all required scheduled follow up visits.

Exclusion Criteria:

1. Subject has a congenital unicuspid or bicuspid aortic valve.
2. Subject with an acute myocardial infarction within 30 days of the index procedure (defined as Q-wave MI or non-Q-wave MI with total CK elevation ≥ twice normal in the presence of CK-MB elevation and/or troponin level elevation).
3. Subject has had a cerebrovascular accident or transient ischemic attack within the past 6 months prior to study enrollment.
4. Subject has end-stage renal disease or has GFR <20 (based on Cockcroft-Gault formula).
5. Subject has a pre-existing prosthetic aortic or mitral valve.
6. Subject has severe (4+) aortic, tricuspid, or mitral regurgitation.
7. Subject has a need for emergency surgery for any reason.
8. Subject has a history of endocarditis within 6 months of index procedure or evidence of an active systemic infection or sepsis.
9. Subject has echocardiographic evidence of new intra-cardiac vegetation or intraventricular or paravalvular thrombus requiring intervention.
10. Subject has Hgb <9 g/dL, platelet count <50,000 cells/mm3 or >700,000 cells/mm3, or white blood cell count <1,000 cells/mm3.
11. Subject requires chronic anticoagulation therapy after the implant procedure and cannot be treated with warfarin (other anticoagulants are not permitted in the first month) for at least 1 month concomitant with either aspirin or clopidogrel.
12. Subject has had a gastrointestinal bleed requiring hospitalization or transfusion within the past 3 months, or has other clinically significant bleeding diathesis or coagulopathy that would preclude treatment with required antiplatelet regimen, or will refuse transfusions.
13. Subject has known hypersensitivity to contrast agents that cannot be adequately pre-medicated, or has known hypersensitivity to aspirin, all P2Y12 inhibitors, heparin, nickel, tantalum, titanium, or polyurethanes.
14. Subject has a life expectancy of less than 12 months due to non-cardiac, comorbid conditions based on the assessment of the investigator at the time of enrollment.
15. Subject has hypertrophic obstructive cardiomyopathy.
16. Subject has any therapeutic invasive cardiac or vascular procedure within 30 days prior to the index procedure (except for balloon aortic valvuloplasty and pacemaker implantation, which are allowed).
17. Subject has untreated coronary artery disease, which in the opinion of the treating physician, is clinically significant and requires revascularization.
18. Subject has severe left ventricular dysfunction with ejection fraction <20%.
19. Subject is in cardiogenic shock or has hemodynamic instability requiring inotropic support or mechanical support devices.
20. Subject has severe vascular disease that would preclude safe access (e.g., aneurysm with thrombus that cannot be crossed safely, marked tortuosity, significant narrowing of the abdominal aorta, severe unfolding of the thoracic aorta, or symptomatic carotid or vertebral disease).
21. Subject has thick (>5 mm) protruding or ulcerated atheroma in the aortic arch.
22. Subject has arterial access that is not acceptable for the LOTUS Edge delivery system and its compatible Lotus Introducer as defined in the Instructions For Use.
23. Subject has current problems with substance abuse (e.g., alcohol, etc.).
24. Subject is participating in another investigational drug or device study that has not reached its primary endpoint.
25. Subject has untreated conduction system disorder (e.g., Type II second degree atrioventricular block) that in the opinion of the treating physician is clinically significant and requires a pacemaker implantation (based on the latest available ESC guidelines). Enrollment is permissible after permanent pacemaker implantation.
26. Subject has severe incapacitating dementia.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-04-01 (Estimated); Primary Completion 2018-10-30 (Estimated); Study Completion 2018-12-30 (Estimated)

PRIMARY OUTCOMES:
Mean aortic valve pressure gradient as measured by echocardiography and assessed by an independent core laboratory. | 30 days post-procedure

IPD SHARING:
Plan to Share IPD: No